CLINICAL TRIAL: NCT02811237
Title: Criteria for Hospitalization or Outpatient Management of Patients With Pulmonary Embolism, Hestia Rule Versus Simplified PESI Score : an Open-label Controlled Randomized International Trial (HOME-PE)
Brief Title: Hospitalization or Out-treatment ManagEment of Patients With Pulmonary Embolism: a Randomized Controlled Trial
Acronym: HOME-PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: European Georges Pompidou Hospital (Other); Hospital Universitario Ramon y Cajal (Other); Leiden University Medical Center (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHRC 2015-04
Record Dates: First submitted 2016-06-07; First posted 2016-06-23 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HESTIA group (Other)
  Interventions: Other: HESTIA
- sPESI group (Other)
  Interventions: Other: sPESI

INTERVENTIONS:
Other: HESTIA — Management based on the HESTIA rule:
  * If the rule is negative, meaning that patient meet none of the exclusion criteria of the rule, the proposed management will be outpatient care.
  * In the other cases, the patient will receive in-hospital care.
  Any reason for management (hospitalization or outpatient treatment) not based on the recommendation will be explained and documented in the e-CRF.
  Arms: HESTIA group
Other: sPESI — Management based on the simplified PESI score:
  * If the sPESI score =0, the proposed management will be outpatient care.
  * In the other cases, the patient will receive in-hospital care.
  Any reason for management (hospitalization or outpatient treatment) not based on the recommendation will be explained and documented in the e-CRF.
  Arms: sPESI group

SUMMARY:
Several studies have demonstrated the possibility of outpatient management or early discharge for certain patients presenting acute pulmonary embolism (PE), providing a suitable structure is in place.

The approach featured in the most recent guidelines on acute PE of the European Society of Cardiology, refers to an all-cause mortality risk assessment using the Pulmonary Embolism Severity Index (PESI) score or the simplified PESI score (sPESI). The sPESI takes into account demographics (age), patient history (cancer, cardiac or respiratory disease), and clinical data (systolic blood pressure, heart rate, oxygen saturation). Outpatient care is offered to low-risk patients, providing that all the conditions pertaining to start anticoagulant treatment and follow-up at home are met.

An alternative approach based on a list of simple criteria has been developed as the one used in HESTIA study. The main criteria included in the HESTIA rule consist of absence of the following: hemodynamic instability, need for oxygen therapy, high-risk of hemorrhage, renal or liver failure, or other medical or social conditions requiring hospitalization.

The investigators hereby propose comparing these two approaches in an open-label, controlled randomized international trial with blinded adjudication of endpoints.

The main objective is to demonstrate, in normotensive PE patients, that a strategy based on the HESTIA rule compared to a strategy based on the simplified PESI score is at least as safe as regards the 30-day-rate of adverse events (recurrent VTE, major bleeding or death).

The major secondary objectives are to demonstrate, in normotensive PE patients, that a strategy based on the HESTIA rule compared to a strategy based on the simplified PESI score is more effective :

* As regards the rate of patients eventually managed as outpatients.
* As regards the rate of patients, in theory, eligible for outpatient care,

DETAILED DESCRIPTION:
All patients admitted in the Emergency Department of the participating centres and diagnosed with PE will be eligible and assessed for potential inclusion.

Included patients will be randomized into two groups (1:1) and stratified by centre. Data will be recorded in a computerized case report form (e-CRF) enabling the randomization.

The HESTIA group will receive outpatient care proposal based on HESTIA criteria. The sPESI group will receive outpatient care proposal based on the simplified PESI score. Any reason for management (hospitalization or outpatient treatment) not based on the recommendation will be explained and documented in the e-CRF.

Follow-up will occur within 72 hours after inclusion, at 14 days, 1 month, and 3 months in both groups to gather clinical event data (recurrent VTE, major bleeding, death), treatment data, unscheduled hospitalizations and patient satisfaction assessment results.

The major objectives will test HESTIA based strategy versus sPESI based strategy in a hierarchical approach:

* step 1: non-inferiority analysis on the rate of adverse events,
* if yes, step 2: superiority analysis on the rate of patients managed as outpatients,
* if yes, step3: superiority analysis on the rate of patients, in theory, eligible for outpatient care.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Emergency Department or unscheduled consultation in one of the participating centres;
* Symptomatic pulmonary embolism objectively confirmed according to the European Society of Cardiology criteria
* Insurance cover according to local legislation;
* Age ≥18 years;
* Free informed consent according to local legislation

Exclusion Criteria:

* Shock or hypotension defined as systolic blood pressure <90 mmHg or a systolic pressure drop by ≥40 mmHg, for >15 minutes, if not caused by new-onset arrhythmia, hypovolaemia, or sepsis;
* Diagnosis of pulmonary embolism established more than 24H before inclusion;
* More than 48h between first presentation to the Emergency unit and inclusion - - Factors rendering 30-day follow-up impossible;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1975 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
The rate of the composite of recurrent VTE, major bleeding and all cause death at 30 days | 30 days
  * Recurrent VTE: objectively confirmed pulmonary embolism or deep venous thrombosis objectively confirmed.
  * Major bleeding: according to the International Society on Thrombosis and Haemostasis' criteria.
  * Death: all-cause mortality.

SECONDARY OUTCOMES:
The rate of patients actually managed as outpatients (meaning patients discharged home within 24 hours after the inclusion in the study (first major secondary objective)) | 1 day
  The rate of patients managed as outpatients defined by patients discharged home within 24 hours after the inclusion in the study.
The rate of "low-risk" patients in theory eligible for outpatient care (second major secondary objective) | 1 day
  The rate of "low-risk" patients eligible for outpatient care:
  * HESTIA group: patients meeting none of the exclusion criteria of the rule (HESTIA rule negative);
  * sPESI group: patients with a simplified PESI score =0.
Safety endpoints - Rate of cumulative events | 14 days, 30 days, 90 days
  The rate of the composite of recurrent VTE, major bleeding and all-cause death,
Safety endpoints - Recurrent VTE | 14 days, 30 days, 90 days
  The rate of recurrent VTE
Safety endpoints - Suspected recurrent VTE | 14 days, 30 days, 90 days
  The rate of recurrent VTE suspicion
Safety endpoints - Major Bleeding | 14 days, 30 days, 90 days
  The rate of major bleeding
Safety endpoints - Non major bleeding | 14 days, 30 days, 90 days
  The rate of non-major clinically relevant bleeding
Safety endpoints - Death | 14 days, 30 days, 90 days
  The rate of all-cause death
Safety endpoints - Serious adverse event | 14 days, 30 days, 90 days
  The rate of serious adverse event as defined in good clinical practice
Applicability of management strategies | 1 day
  The rate of patients actually managed as outpatients among number of patientpatients eligible for outpatient management
Resources utilization | Day 90
  Resources utilization will be assessed via the cumulative in-hospital length of stay (LOS) defined as the LOS for initial hospitalization plus LOS of possible unscheduled hospitalizations in the 30 days and 3 months following admission.
Patient satisfaction with care | 30 days
  A specific questionnaire will be used at 30 days following inclusion:
  - Anti-Clot Treatment - Specific Questionnaire (ACTS)
Patient quality of life | 30 days
  A specific questionnaire will be used at 30 days following inclusion:
  - Patient-reported Pulmonary Embolism Quality of Life Questionnaire (PEmb-QoL).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie ROY, MD.PhD, Principal Investigator — CHU d'Angers, France; Olivier SANCHEZ, MD.PhD, Principal Investigator — APHP Hôpital Européen Georges Pompidou, Paris, France; Menno HUISMAN, MD.PhD, Principal Investigator — Leiden University Medical Center, Leiden, The Netherlands; David JIMENEZ, MD.PhD, Principal Investigator — Hospital Universitario Ramon y Cajal, Madrid, Spain; Andréa PENALOZA, MD.PhD, Principal Investigator — Clinique Unisersitaire Saint Luc, Brussels, Belgium; Guy MEYER, MD.PhD, Study Chair — APHP Hôpital Européen Georges Pompidou, Paris, France; EriK KLOK, MD, Principal Investigator — Leiden University Medical Center Leiden, the Netherlands; Olivier HUGLI, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (28):
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hôpital Erasme, Brussels
  - Hôpital Saint-Pierre, Brussels
  - CHU de Liège, Liège
  - Hôpital de Namur, Namur
- France (16):
  - Angers University Hospital, Angers
  - Hia Brest, Brest
  - CHU Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - APHP Louis Mourier, Colombes
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Thibault Schotté, Le Mans
  - CHU de Montpellier, Montpellier
  - APHP Cochin, Paris
  - APHP Hôpital Européen Georges Pompidou, Paris
  - APHP Lariboisière, Paris
  - CHU de Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CH Toulon, Toulon
  - CHU Toulouse, Toulouse
- Netherlands (4):
  - Red Cross Hospital, Beverwijk
  - TERGOOI, Hilversum
  - Leiden University Medical Center Leiden,, Leiden
  - University Medical Center Utrecht, Utrecht
- Ramon y Cajal Hospital, Madrid, Spain
- Switzerland (2):
  - Hôpital de Genève, Geneva
  - Hôpital de Lausanne, Lausanne

REFERENCES:
- [Background] Piran S, Le Gal G, Wells PS, Gandara E, Righini M, Rodger MA, Carrier M. Outpatient treatment of symptomatic pulmonary embolism: a systematic review and meta-analysis. Thromb Res. 2013 Nov;132(5):515-9. doi: 10.1016/j.thromres.2013.08.012. Epub 2013 Aug 28. PMID 24035045
- [Background] Zondag W, Kooiman J, Klok FA, Dekkers OM, Huisman MV. Outpatient versus inpatient treatment in patients with pulmonary embolism: a meta-analysis. Eur Respir J. 2013 Jul;42(1):134-44. doi: 10.1183/09031936.00093712. Epub 2012 Oct 25. PMID 23100493
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Aujesky D, Roy PM, Verschuren F, Righini M, Osterwalder J, Egloff M, Renaud B, Verhamme P, Stone RA, Legall C, Sanchez O, Pugh NA, N'gako A, Cornuz J, Hugli O, Beer HJ, Perrier A, Fine MJ, Yealy DM. Outpatient versus inpatient treatment for patients with acute pulmonary embolism: an international, open-label, randomised, non-inferiority trial. Lancet. 2011 Jul 2;378(9785):41-8. doi: 10.1016/S0140-6736(11)60824-6. Epub 2011 Jun 22. PMID 21703676
- [Background] Zondag W, Mos IC, Creemers-Schild D, Hoogerbrugge AD, Dekkers OM, Dolsma J, Eijsvogel M, Faber LM, Hofstee HM, Hovens MM, Jonkers GJ, van Kralingen KW, Kruip MJ, Vlasveld T, de Vreede MJ, Huisman MV; Hestia Study Investigators. Outpatient treatment in patients with acute pulmonary embolism: the Hestia Study. J Thromb Haemost. 2011 Aug;9(8):1500-7. doi: 10.1111/j.1538-7836.2011.04388.x. PMID 21645235
- [Derived] Roy PM, Penaloza A, Hugli O, Klok FA, Arnoux A, Elias A, Couturaud F, Joly LM, Lopez R, Faber LM, Daoud-Elias M, Planquette B, Bokobza J, Viglino D, Schmidt J, Juchet H, Mahe I, Mulder F, Bartiaux M, Cren R, Moumneh T, Quere I, Falvo N, Montaclair K, Douillet D, Steinier C, Hendriks SV, Benhamou Y, Szwebel TA, Pernod G, Dublanchet N, Lapebie FX, Javaud N, Ghuysen A, Sebbane M, Chatellier G, Meyer G, Jimenez D, Huisman MV, Sanchez O; HOME-PE Study Group. Triaging acute pulmonary embolism for home treatment by Hestia or simplified PESI criteria: the HOME-PE randomized trial. Eur Heart J. 2021 Aug 31;42(33):3146-3157. doi: 10.1093/eurheartj/ehab373. PMID 34363386